CLINICAL TRIAL: NCT04910516
Title: Examining the Effect of "Emotional Freedom Technique" on Covid-19 Reasoned Fear and Anxiety Levels of Nurses Working in the Emergency Department
Brief Title: Emotional Freedom Technique (EFT) Effect on Nurses
Acronym: EFT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Marmara University (Other)
Responsible Party: Principal Investigator, gulsah okut, Principal Investigator, Marmara University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: B.10.1.TKH.4.34.H.GP.0.01/120
Record Dates: First submitted 2021-05-27; First posted 2021-06-02 (Actual); Last update posted 2021-06-02 (Actual); Status verified 2021-05

CONDITIONS: Anxiety, Covid-19 Fear
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: It was aimed to measure the anxiety and covid-19 fears of the Emergency Department nurses. The number of people to be included in the study was determined to be working with 44 nurses in the experimental group and 44 nurses in the control group in the calculation made for a maximum 5% type I error and at least 80% power. The determination of the sample size and the creation of the Randomization Table was calculated using the "www.e-picos.com", NY New York, program.
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (No Intervention): The nurses in the control group were informed about the purpose of working in a quiet room. STAI-D, STAI-S, SUD, P19-S scales were filled face-to-face by the investigator after their informed consent was obtained. The scales were filled again by the researcher after a break of 7 (seven) days.
- Experiment Group (Experimental): In order to avoid bias in the intervention applied in our study, the experimental group was started after the control group was finished. The participants were informed about the purpose of working face-to-face in a quiet room so that EFT, which will be applied online for 7 (seven) days by the researcher, can be applied effectively and accurately. STAI-D, STAI-S, SUD, P19-S scales were completed after their consent was obtained. The researcher, who has the EFT certificate, first showed the application steps on himself with the guidance of the EFT guideline, and ensured that the application steps were applied again simultaneously on both himself and the participant. After this application, it was provided to make EFT online for 7 (seven) days. STAI-D, STAI-S, SUD, P19-S scales were filled in after the last EFT application.
  Interventions: Behavioral: Emotional Freedom Techniques (EFT)

INTERVENTIONS:
Behavioral: Emotional Freedom Techniques (EFT) — It combines cognitive therapy, acceptance and stability therapy, and acupuncture point stimulation, and is based on manual stimulation of acupuncture points specific to Shiatsu or other acupressure massage fo
  Arms: Experiment Group

SUMMARY:
It has been planned to determine the effect of EFT, which effectiveness has been determined by the studies, on the covid-19 fear and anxiety experienced by the nurses working in the emergency department. The study was designed as a randomized controlled study with pre-test and post-test control group.

DETAILED DESCRIPTION:
Although it has been a year since WHO declared an emergency, the covid-19 virus has mutated and the number of cases has started to increase again as of February 2021. The emergence of uncertainties in the risk of transmission of the mutant virus together with the simultaneous management of both the care process of pandemic patients and the patients who apply for emergency care and treatment in the emergency services increases the fear of the virus. The feeling of fear causes the person to become distracted and increase anxiety by focusing on the fact that he or she is under the threat of the virus. Recently, non-pharmacological techniques are widely used to reduce anxiety and fear. One of them is EFT. It is to examine the effects of EFT, which effectiveness has been determined with the studies carried out in this challenging process, on the covid-19 fear and high anxiety of emergency room nurses.

ELIGIBILITY:
Inclusion Criteria:

* Not taking any courses about coping with anxiety and stress,
* Volunteering to participate in the study,
* The absence of infection, wound, scar in the tapping area

Exclusion Criteria:

* Having any psychiatric diagnoses

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 88 (Estimated)
Dates: Start 2021-04-10 (Actual); Primary Completion 2021-05-25 (Actual); Study Completion 2021-07-01 (Estimated)

PRIMARY OUTCOMES:
The subjective units of distress scale | After 7 days of EFT
  The cognitive element of EFT involves self-rating of distress severity and pairing of an abbreviated exposure statement and a self-acceptance statement. The severity of distress was evaluated by subjects on an 11-point Likert scale. 0 corresponds to absolutely no distress, while 10 corresponds to the maximum possible distress. This was considered as the subjective units of distress scale (SUD) and provides clinicians and patients with the measurement of the severity of symptoms experienced by the latter in addition to a repeated measure by which the progress can be evaluated.
State-Trait Anxiety Inventory | After 7 days of EFT
  This scale consists of a total of forty items; the "State Anxiety Scale" consisting of twenty items and the "Trait Anxiety Scale" consisting of twenty items. There are two types of expressions in the scales: direct and reversed. Direct expressions express negative emotions, and reversed expressions express positive emotions. There are ten (1, 2, 5, 8, 10, 11, 15, 16, 19, and 20th) reversed statements on the state anxiety scale. On the trait anxiety scale, there are seven (1, 6, 7, 10, 13, 16, 19th items) reversed. The total score value obtained from each scale is between minimum 20 and maximum 80. The total score of the reverse expressions is subtracted from the total score obtained for direct expressions. A predetermined and constant value is added to this number. This is 50 for state anxiety and 35 for trait anxiety. The most recent value is the individual's anxiety score. A high score indicates a high anxiety level, a small score indicates a low anxiety level.
Coronavirus-19 Fear Scale | After 7 days of EFT
  This scale consists of 7 items in total and is collected in one dimension.There are no reverse questions in the scale and are answered in a five-point Likert type (1 = Strongly disagree, 5 = Strongly agree).The minimum score that can be obtained for each question on the scale is 1, and the maximum score is 5. The total score that can be obtained from the scale varies between 7-35. As the total score on the scale increases, the fear of coronavirus increases

CONTACTS AND LOCATIONS:
Locations (1):
- Marmara University, Istanbul, Kadikoy, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Sun N, Wei L, Shi S, Jiao D, Song R, Ma L, Wang H, Wang C, Wang Z, You Y, Liu S, Wang H. A qualitative study on the psychological experience of caregivers of COVID-19 patients. Am J Infect Control. 2020 Jun;48(6):592-598. doi: 10.1016/j.ajic.2020.03.018. Epub 2020 Apr 8. PMID 32334904
- [Background] Clond M. Emotional Freedom Techniques for Anxiety: A Systematic Review With Meta-analysis. J Nerv Ment Dis. 2016 May;204(5):388-95. doi: 10.1097/NMD.0000000000000483. PMID 26894319